CLINICAL TRIAL: NCT03589768
Title: A Phase II Double-Blind Trial to Evaluate the Safety, Immunogenicity and Effect on Infant Immune Responses of a Single Dose of Tdap in Pregnant Women in Mali
Brief Title: Study on the Safety and Immunogenicity of Boostrix Vaccine in Pregnant Malian Women and Their Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0024
Record Dates: First submitted 2018-06-14; First posted 2018-07-18 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2018-10-04

CONDITIONS: Clostridium Difficile Immunisation; Diphtheria; Diphtheria Immunisation; Pertussis; Tetanus; Tetanus Immunisation
Keywords: BOOSTRIX; Immunogenicity; Infant; Mali; Phase II; Pregnant Women; Safety; Tdap
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): 0.5 ml single dose of Tdap (Tetanus, Diphtheria, Acellular Pertussis Vaccine), BOOSTRIX administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated Gestational Age (GA).
  N=133
  Interventions: Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed onto aluminum hydroxide
- Group 2 (Active Comparator): 0.5 ml single dose of Td (Tetanus, Diphtheria Toxoid) administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated GA.
  N=67
  Interventions: Biological: Tetanus and Diphtheria Toxoids Adsorbed

INTERVENTIONS:
Biological: Tetanus and Diphtheria Toxoids Adsorbed — Used for active immunization of adults and children 7 years of age and older against diphtheria and tetanus.
  Arms: Group 2
Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed onto aluminum hydroxide — A sterile isotonic suspension of tetanus and diphtheria toxoids and pertussis antigens adsorbed on Aluminum hydroxide.
  Arms: Group 1

SUMMARY:
This is a phase II, randomized, double-blind, active-controlled study to evaluate the safety, immunogenicity, and effect on infant immune responses of a single dose of Tetanus diphtheria acellular pertussis vaccine (Tdap) in pregnant women in Mali. 200 healthy pregnant women, ages 18 through 39 years, inclusive, who meet all eligibility criteria will be randomly allocated in a 2:1 ratio to receive either Tdap (BOOSTRIX) or Tetanus diphtheria toxoid (Td) at 14 0/7 weeks through 26 6/7 weeks estimated Gestational Age (GA). For the fetuses of pregnant subjects, GA will be established by ultrasound, whenever possible, in combination with date of last menstrual period (LMP), when available, and fundal height. Study duration is 21 months: approximately 2 months in the start-up period, 6 months enrolling subjects, and 13 months (3-7 months while pregnant and 6 months postpartum) from last subject vaccinated until she and her infant complete follow-up. The primary objectives of this study are: 1) to assess the safety and tolerability of a single 0.5 mL intramuscular injection of BOOSTRIX in pregnant women; 2) to assess the safety of a single maternal BOOSTRIX vaccination on the fetus and infant; 3) to assess the level of Pertussis Toxin (PT) antibody at birth among infants whose mothers received a single dose of BOOSTRIX or Td while pregnant.

DETAILED DESCRIPTION:
This is a phase II, randomized, double-blind, active-controlled study to evaluate the safety, immunogenicity, and effect on infant immune responses of a single dose of Tetanus diphtheria acellular pertussis vaccine (Tdap) in pregnant women in Mali. 200 healthy pregnant women, ages 18 through 39 years, inclusive, who meet all eligibility criteria will be randomly allocated in a 2:1 ratio to receive either Tdap (BOOSTRIX) or Tetanus diphtheria toxoid (Td) at 14 0/7 weeks through 26 6/7 weeks estimated Gestational Age (GA). For the fetuses of pregnant subjects, GA will be established by ultrasound, whenever possible, in combination with date of last menstrual period (LMP), when available, and fundal height. Study duration is 21 months: approximately 2 months in the start-up period, 6 months enrolling subjects, and 13 months (3-7 months while pregnant and 6 months postpartum) from last subject vaccinated until she and her infant complete follow-up. The primary objectives of this study are: 1) to assess the safety and tolerability of a single 0.5 mL intramuscular injection of BOOSTRIX in pregnant women; 2) to assess the safety of a single maternal BOOSTRIX vaccination on the fetus and infant; 3) to assess the level of Pertussis Toxin (PT) antibody at birth among infants whose mothers received a single dose of BOOSTRIX or Td while pregnant. The secondary objectives are: 1) to assess the antibody response to BOOSTRIX vaccine antigens in pregnant women one month after receipt of BOOSTRIX, at the time of delivery, and at 6 months after delivery; 2) to compare the antibody levels of BOOSTRIX vaccine antigens at birth (cord blood) and 6 weeks of age (before receiving any infant doses of Diphtheria, Tetanus, and whole-cell Pertussis (DTwP)) in infants whose mothers received BOOSTRIX or Td during pregnancy; 3) to assess placental antibody transfer by determining the ratio of maternal and infant BOOSTRIX -specific antibody responses at delivery; 4) to assess interference with infant antibody responses to DTwP either prior to the second dose of the primary DTwP series, at approximately 10 weeks of age (in 1/2 of subjects), or approximately one month after the third dose of the primary DTwP series, at approximately 18 weeks of age (in 1/2 of subjects), and at 6 months of age (all subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant woman 18-39 years of age, inclusive.
2. Singleton fetus, with estimated gestational age of 14 0/7 through 26 6/7 weeks gestation, inclusive, on the day of study vaccination.
3. Provide written consent after the nature of the study has been explained according to local regulatory requirements and prior to any study procedures*.

   *Prior to obtaining individual informed consent for each subject, the investigators will obtain community consent by discussing the trial with all the appropriate local groups, as necessary, to obtain permission to approach the subjects. Written, informed consent for participation in the trial will be obtained by the investigators from all individual subjects. The consent forms will be written in French, the official language of Mali, and will be translated into Bambara, the most prevalent of the local languages, and recorded on audiotape.
4. In good health as determined by medical history, targeted physical examination* (physical examination performed as part of routine antenatal care of a study-specific brief exam may be used to determine eligibility), vital signs (oral temperature < 37.8 degrees Celsius; pulse 55 to 100 beats per minute (bpm), inclusive; systolic blood pressure 90 to 140 millimeters of mercury (mm Hg), inclusive; diastolic blood pressure 55 to 90 mm Hg, inclusive), and clinical judgment of the investigator.

   *If indicated based on medical history, to evaluate acute or currently ongoing chronic medical diagnoses or conditions that would affect the assessment of eligibility and safety of subjects. Chronic medical diagnoses or conditions being actively managed must be within acceptable limits in the last 180 days. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and the study vaccination are acceptable provided the subject is asymptomatic, condition stable, and there is no additional risk to the subject or interference with the evaluation of responses to the study vaccination.
5. Ability to comprehend and comply with all study procedures, as determined by the investigator determining eligibility, and availability for follow-up.
6. Willing to allow study staff to gather pertinent medical information, including pregnancy outcome data and medical information about her infant.

Exclusion Criteria:

1. History of illness or an ongoing illness that, in the opinion of the investigator, may pose additional risk to the subject or her fetus if she participates in the study.
2. Infection requiring systemic antibiotics or antiviral treatment within the 7 days prior to study vaccination.
3. Fever (oral temperature > / = 37.8 degrees Celsius/100.0 degrees Fahrenheit) or other acute illness within 3 days prior to study vaccination*.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
4. Known active neoplastic disease (excluding non-melanoma skin cancer), anticancer chemotherapy, or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. History of any hematologic malignancy at any time.
6. A history of a serious adverse event following previous immunizations (e.g., Bell's Palsy, Guillain-Barre Syndrome, encephalopathy), or history of progressive neurologic disorders.
7. Known or suspected disease that impairs the immune system including known or suspected HIV infection or HIV-related disease.
8. Receipt of immunosuppressive therapy, including long-term use of glucocorticoids: oral, inhaled, intranasal or parenteral prednisone > / = 20 mg/day or equivalent for more than 2 weeks within the 30 days prior to enrollment. Use of topical corticosteroids is allowed.
9. Known hepatitis B or hepatitis C infection, by history or medical record.
10. Behavioral or cognitive impairment or psychiatric disease (includes hospitalization for psychiatric illness, suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination) that, in the opinion of the investigator, may interfere with the subject's ability to participate in the trial.
11. Have a history of alcohol or drug abuse within 5 years prior to study vaccination (that is believed by the site investigator to potentially interfere with the subject's ability to participate in the study).
12. Known hypersensitivity or allergy to any component of the study vaccine (formaldehyde, alum).
13. History of severe allergic reaction (e.g., anaphylaxis) after a previous dose of BOOSTRIX or any other vaccine directed against tetanus, diphtheria, or pertussis.
14. Receipt or planned receipt of any live licensed vaccine within 30 days before or after vaccination or any inactivated licensed vaccine within 14 days before or after vaccination.
15. Receipt of immunoglobulin (except RhoGAM, which is allowed) or other blood products within 90 days prior to study vaccination.
16. Receipt of an experimental agent or device within 30 days prior to vaccination, or the expected receipt of an experimental agent* (other than BOOSTRIX) during this trial-reporting period.

    *Experimental agents include vaccines, drugs, biologics, devices, blood products, and medications. Subjects who have received a licensed product, as a subject in a clinical trial, within 30 days prior to vaccination or who are expecting to enroll in such a trial during the study period will also be excluded. Observational studies, surveys, and other studies that do not involve experimental agents or devices are allowed.
17. High risk for serious obstetrical complication (refer to ACOG Practice Bulletins for definitions, as necessary)*.

    *Including the following: (a) gestational hypertension (well controlled history of essential or gestational hypertension, as evidenced by normal BPs as defined above, is allowed), (b) gestational diabetes not controlled by diet and exercise (the use of insulin or glyburide to control gDM, at the time of enrollment, is exclusionary), (c) current pre-eclampsia or eclampsia, (d) known current multiple gestation, (e)history of preterm delivery before EGA 35 weeks 0 days or current preterm labor, and/or (f) known intrauterine fetal growth restriction (defined as ultrasound confirmation of an estimated fetal weight that is less than the 10th percentile for gestational age).
18. Pregnant with a fetus with a known or suspected major congenital anomaly or genetic abnormality.
19. Study personnel or immediate family members (brother, sister, child, parent) or the spouse of study personnel.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 399 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States
- Center for Vaccine Development - Mali, Bamako, Mali

REFERENCES:
- [Derived] Haidara FC, Tapia MD, Diallo F, Portillo S, Williams M, Traore A, Rotrosen E, Hensel E, Makowski M, Selamawi S, Powell JA, Kotloff KL, Pasetti MF, Sow SO, Neuzil KM. Safety and immunogenicity of a single dose of Tdap compared to Td in pregnant women in Mali and 3 its effect on infant immune responses: a single-centre, randomised, double-blind, active-controlled phase 2 study. EClinicalMedicine. 2024 Mar 28;71:102556. doi: 10.1016/j.eclinm.2024.102556. eCollection 2024 May. PMID 38586589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for this study include pregnant women in their first and second trimesters, 18 to 39 years of age, inclusive, who met all eligibility criteria and were deemed to be in good health. The infants of the pregnant participants were also enrolled and followed from birth to 6 months of age. Participants were enrolled between 24JAN2019 and 03JAN2020.
Groups:
- BOOSTRIX - Maternal: 0.5 ml single dose of Tdap (Tetanus, Diphtheria, Acellular Pertussis Vaccine), BOOSTRIX administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated Gestational Age (GA).
  Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed onto aluminum hydroxide: A sterile isotonic suspension of tetanus and diphtheria toxoids and pertussis antigens adsorbed on Aluminum hydroxide.
- Td - Maternal; Td - Infant: 0.5 ml single dose of Td (Tetanus, Diphtheria Toxoid) administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated GA.
  Tetanus and Diphtheria Toxoids Adsorbed: Used for active immunization of adults and children 7 years of age and older against diphtheria and tetanus.
- BOOSTRIX - Infant: 0.5 ml single dose of Tdap (Tetanus, Diphtheria, Acellular Pertussis Vaccine), BOOSTRIX administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated GA.
  Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed onto aluminum hydroxide: A sterile isotonic suspension of tetanus and diphtheria toxoids and pertussis antigens adsorbed on Aluminum hydroxide.
Period: Overall Study
Arm/Group | BOOSTRIX - Maternal | Td - Maternal | BOOSTRIX - Infant | Td - Infant
Started | 134 | 67 | 131 | 67
Completed | 130 | 67 | 123 | 64
Not Completed | 4 | 0 | 8 | 3
Not completed — Death | 1 | 0 | 8 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all maternal participants who received the study vaccine or infants born to mothers who received the study vaccine.
Groups:
- BOOSTRIX - Maternal: 0.5 ml single dose of Tdap, BOOSTRIX administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated Gestational Age (GA).
- Td - Maternal: 0.5 ml single dose of Td administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated GA.
- BOOSTRIX - Infant: Infants of pregnant women who received 0.5 ml single dose of Tdap, BOOSTRIX administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated Gestational Age (GA).
- Td - Infant: Infants of pregnant women who received 0.5 ml single dose of Td administered intramuscularly to pregnant women at 14 0/7 weeks through 26 6/7 weeks estimated GA.
- Total: Total of all reporting groups
Arm/Group | BOOSTRIX - Maternal | Td - Maternal | BOOSTRIX - Infant | Td - Infant | Total
Number analyzed (Participants) | 133 | 67 | 126 | 66 | 392
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 126 | 66 | 192
  Between 18 and 65 years | 133 | 67 | 0 | 0 | 200
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Ages for each group are represented on separate rows for Mothers and Infants. Infants were enrolled in the study upon birth.
  years
    Mothers: number analyzed (Participants) | 133 | 67 | 0 | 0 | 200
    Mothers | 25.7 (5.6) | 25.4 (5.4) |  |  | 25.6 (5.5)
    Infants: number analyzed (Participants) | 0 | 0 | 126 | 66 | 192
    Infants |  |  | 0 (0) | 0 (0) | 0 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 67 | 58 | 34 | 292
  Male | 0 | 0 | 68 | 32 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 133 | 67 | 126 | 66 | 392
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 133 | 67 | 126 | 66 | 392
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mali | 133 | 67 | 126 | 66 | 392
Gestational Age (GA) at Vaccination (weeks) [Count of Participants; unit: Participants] — GA available for maternal participants only. Population: Gestational Age at Vaccination is only available for participants in the Maternal groups.
  Participants
    14-17 weeks: number analyzed (Participants) | 133 | 67 | 0 | 0 | 200
    14-17 weeks | 58 | 35 |  |  | 93
    18-21 weeks: number analyzed (Participants) | 133 | 67 | 0 | 0 | 200
    18-21 weeks | 42 | 12 |  |  | 54
    22-26 weeks: number analyzed (Participants) | 133 | 67 | 0 | 0 | 200
    22-26 weeks | 33 | 20 |  |  | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Pregnant Women Reporting Related Serious Adverse Events (SAEs) and Unrelated SAEs
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. All SAEs were reported from time of first study vaccination through approximately 6 months after the first study vaccination
Time Frame: Study Day 1 through Day 180 (6-months post-partum)
Population: The maternal safety analysis population includes all pregnant women who received the study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 133 | 67
Participants
  Related SAEs | 0 | 0
  Unrelated SAEs | 20 | 10
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Test type: Other — N/A, Only risk difference estimated and 95% CI reported; Risk Difference (RD) = 0.1, 95% CI 2-sided [-11.9 to 10.3] — Difference is calculated as the proportion in the BOOSTRIX group minus the proportion in the Td group

2. Primary Outcome: Number of Pregnant Women Reporting Pregnancy-Specific Adverse Events (AEs)
Description: Pregnancy related AEs include: pregnancy loss (graded as severe [grade 3] if occurred), bleeding during pregnancy prior to the onset of labor, postpartum hemorrhage, postabortal endometritis/salpingitis, preterm rupture of membranes, preterm contractions/labor/delivery, poor fetal growth, hypertension, preeclampsia/eclampsia, chorioamnionitis, postpartum endometriosis, gestational diabetes mellitus, and/or pregnancy-related clinical AE not previously identified in this list.
Time Frame: Study Day 1 through Day 180 (6-months post-partum)
Population: The maternal safety analysis population includes all pregnant women who received the study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 133 | 67
Participants
  Mild AEs | 5 | 1
  Moderate AEs | 8 | 7
  Severe AEs | 13 | 5
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Test type: Superiority; p = 0.559, Fisher Exact; Risk Difference (RD) = 4.62, 95% CI 2-sided [-6.25 to 15.5] — Difference is calculated as the proportion in the BOOSTRIX group minus the proportion in the Td group

3. Primary Outcome: Number of Infants Reporting Related SAEs and Unrelated SAEs
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. All SAEs were reported from time of birth through 6 months of age.
Time Frame: Birth Day through 6 months of age
Population: The infant safety analysis population includes all infants born during the study via live birth to women who received the study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 126 | 66
Participants
  Related SAEs | 0 | 0
  Unrelated SAEs | 13 | 6
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Test type: Other — Only risk difference estimated and 95% CI reported; Risk Difference (RD) = 1.2, 95% CI 2-sided [-9.3 to 9.8]; Difference is calculated as the proportion in the BOOSTRIX group minus the proportion in the Td group

4. Primary Outcome: Number of Infants Reporting Pregnancy-specific AEs
Description: Infant pregnant related AEs include: preterm birth, low birth weight, neonatal complications in a term infant, congenital anomalies/birth defects, and/or clinical AE in the newborn not identified previously in this list.
Time Frame: Birth Day through 6 months of age
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 126 | 66
Participants
  Mild AEs | 0 | 0
  Moderate AEs | 15 | 5
  Severe AEs | 6 | 2
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Test type: Superiority; p = 0.290, Fisher Exact; Risk Difference (RD) = 6.06, 95% CI 2-sided [-3.82 to 15.9]; Difference is calculated as the proportion in the BOOSTRIX group minus the proportion in the Td group

5. Primary Outcome: Number of Pregnant Women Reporting Solicited Injection Site and Systemic Reactogenicity Events
Description: Local AEs solicited on a memory aid provided to participants included Pain, Tenderness, Ecchymosis (functional grade based on interference with daily activities), Ecchymosis (any measured value >0mm), Erythema (functional grade), Erythema (any measured value >0mm), Induration (functional grade), and Induration (any measured value >0mm). Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, Allergic reaction, and Nausea. Participants are considered reporting the local or systemic AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Pre-Dose Day 1, Post-Dose Day 1, Day 4, Day 8
Population: The Safety Analysis population includes all pregnant women who received the study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 133 | 67
Participants
  Pre-Dose | 0 | 0
  Post-dose | 3 | 4
  Day 4 | 6 | 8
  Day 8 | 0 | 0

6. Primary Outcome: Number of Pregnant Women Reporting Unsolicited Non-serious AEs
Description: Frequency of all unsolicited non-serious AEs from day of study vaccination (Day 1) to Day 31, compared between those who received BOOSTRIX and those who received Td.
Time Frame: Day 1 through Day 31
Population: The maternal safety analysis population includes all pregnant women who received the study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 133 | 67
Participants | 6 | 2
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Test type: Other — Only risk difference estimated and 95% CI reported; Risk Difference (RD) = 1.5, 95% CI 2-sided [-6.4 to 7.3]; Difference is calculated as the proportion in the BOOSTRIX group minus the proportion in the Td group

7. Primary Outcome: Geometric Mean Concentration (GMC) of Serum IgG Antibodies to Pertussis Toxin (PT) in Infants Born to Women Receiving BOOSTRIX or Td
Description: Geometric Mean Concentration (GMC) of serum IgG antibodies to PT as measured by Enzyme-Linked Immunosorbent Assay (ELISA) at birth between infants born to women vaccinated with BOOSTRIX or Td. DTwP is Diphtheria, Tetanus, and whole cell Pertussis vaccine.
Time Frame: Birth Day, Prior to receipt of first dose of DTwP (approximately 6 weeks of age), One month after receipt of first dose of DTwP (approximately 10 weeks of age), One month after receipt of last dose of DTwP (approximately 18 weeks of age), 6 months of age
Population: The infant mITT population for immunogenicity analyses includes all infants born via live birth to women who received the study vaccination and have a perinatal blood sample for which valid immunogenicity results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 124 | 64
IU/mL
  At birth | 55.4 [46.2 to 66.6] | 7.9 [5.4 to 11.5]
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age): number analyzed (Participants) | 114 | 59
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age) | 21.0 [17.3 to 25.5] | 4.3 [3.0 to 6.2]
  One month after receipt of first dose of DTwP (approximately 10 weeks of age): number analyzed (Participants) | 58 | 32
  One month after receipt of first dose of DTwP (approximately 10 weeks of age) | 15.0 [11.4 to 19.7] | 5.1 [3.3 to 8.1]
  One month after receipt of last dose of DTwP (approximately 18 weeks of age): number analyzed (Participants) | 50 | 25
  One month after receipt of last dose of DTwP (approximately 18 weeks of age) | 20.2 [13.7 to 29.9] | 77.2 [32.2 to 184.8]
  6 months of age: number analyzed (Participants) | 63 | 32
  6 months of age | 17.3 [12.8 to 23.4] | 67.1 [35.5 to 126.7]
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for birth day timepoint; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 7.0, 95% CI 2-sided [4.6 to 10.7] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for Prior to receipt of first dose of DTwP (approximately 6 weeks of age) timepoint; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 4.8, 95% CI 2-sided [3.2 to 7.3] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for One month after receipt of first dose of DTwP (approximately 10 weeks of age) timepoint; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 2.9, 95% CI 2-sided [1.8 to 4.8] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for One month after receipt of last dose of DTwP (approximately 18 weeks of age) time point; Test type: Superiority; p = 0.0068, t-test, 2 sided; Test compares difference in log values; Ratio = 0.3, 95% CI 2-sided [0.1 to 0.7] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 5: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for 6 months of age time point; Test type: Superiority; p = 0.0003, t-test, 2 sided; Test compares differences in log values; Ratio = 0.3, 95% CI 2-sided [0.1 to 0.5] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

8. Secondary Outcome: GMC of Serum IgG Antibodies to PT in Pregnant Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to PT as measured by Enzyme-Linked Immunosorbent Assay (ELISA) between women vaccinated with BOOSTRIX or Td.
Time Frame: Pre-dose Day 1, One month after vaccination, at delivery, Day 180 (approximately 6 months after delivery)
Population: The maternal mITT population for immunogenicity analyses includes all pregnant women who received the study vaccination, have valid immunogenicity results (from blood or breastmilk) at baseline, and at least one post-vaccination visit.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 130 | 66
IU/mL
  Pre-vaccination | 9.1 [7.5 to 11.1] | 9.8 [7.3 to 13.1]
  One month after vaccination: number analyzed (Participants) | 129 | 66
  One month after vaccination | 90.0 [76.8 to 105.6] | 10.4 [7.8 to 13.9]
  Delivery: number analyzed (Participants) | 127 | 64
  Delivery | 47.0 [40.1 to 55.1] | 10.1 [7.4 to 13.6]
  6 months after delivery: number analyzed (Participants) | 65 | 33
  6 months after delivery | 40.9 [33.3 to 50.2] | 12.2 [8.2 to 18.2]
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for pre-vaccination time point; Test type: Superiority; p = 0.7102, t-test, 2 sided; Test compares difference in log values; Ratio = 0.9, 95% CI 2-sided [0.7 to 1.3] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for one month after vaccination time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 8.7, 95% CI 2-sided [6.2 to 12.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for delivery time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 4.7, 95% CI 2-sided [3.3 to 6.6] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for 6 months after delivery time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 3.3, 95% CI 2-sided [2.1 to 5.2] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

9. Secondary Outcome: GMC of Serum IgG Antibodies to Filamentous Hemagglutinin (FHA) in Pregnant Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to FHA as measured by Enzyme-Linked Immunosorbent Assay (ELISA) between women vaccinated with BOOSTRIX or Td.
Time Frame: Pre-dose Day 1, One month after vaccination, at delivery, Day 180 (approximately 6 months after delivery)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 130 | 66
IU/mL
  Pre-vaccination | 28.6 [24.4 to 33.6] | 27.1 [21.5 to 34.2]
  One month after vaccination: number analyzed (Participants) | 129 | 66
  One month after vaccination | 545.3 [463.6 to 641.4] | 29.5 [23.7 to 36.8]
  Delivery: number analyzed (Participants) | 127 | 64
  Delivery | 321.5 [275.0 to 375.8] | 30.6 [24.8 to 37.7]
  6 months after delivery: number analyzed (Participants) | 65 | 33
  6 months after delivery | 259.0 [205.3 to 326.6] | 34.9 [24.7 to 49.3]
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for pre-vaccination time point; Test type: Superiority; p = 0.7039, t-test, 2 sided; Test compares difference in log values; Ratio = 1.1, 95% CI 2-sided [0.8 to 1.4] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for one month after vaccination time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 18.5, 95% CI 2-sided [14.0 to 24.3] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for delivery time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 10.5, 95% CI 2-sided [8.1 to 13.7] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for 6 months after delivery time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Difference in log values back transformed into ratio; Ratio = 7.4, 95% CI 2-sided [5.0 to 11.1]; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

10. Secondary Outcome: GMC of Serum IgG Antibodies to Pertactin (PRN) in Pregnant Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to PRN as measured by Enzyme-Linked Immunosorbent Assay (ELISA) between women vaccinated with BOOSTRIX or Td.
Time Frame: Pre-dose Day 1, One month after vaccination, at delivery, Day 180 (approximately 6 months after delivery)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 130 | 66
IU/mL
  Pre-vaccination | 5.6 [4.4 to 6.9] | 4.6 [3.5 to 6.0]
  One month after vaccination: number analyzed (Participants) | 129 | 66
  One month after vaccination | 255.3 [186.4 to 349.9] | 4.7 [3.6 to 6.2]
  Delivery: number analyzed (Participants) | 127 | 64
  Delivery | 164.6 [121.0 to 224.1] | 5.1 [3.7 to 7.1]
  6 months after delivery: number analyzed (Participants) | 65 | 33
  6 months after delivery | 97.1 [61.5 to 153.5] | 5.1 [3.5 to 7.6]
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for pre-vaccination time point; Test type: Superiority; p = 0.2897, t-test, 2 sided; Test compares difference in log values; Ratio = 1.2, 95% CI 2-sided [0.8 to 1.8] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for one month after vaccination time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 54.2, 95% CI 2-sided [35.6 to 82.4] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for delivery time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 32.0, 95% CI 2-sided [20.6 to 49.7] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for 6 months after delivery time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 18.9, 95% CI 2-sided [10.4 to 34.2] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

11. Secondary Outcome: GMC of Serum IgG Antibodies to Tetanus in Pregnant Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to Tetanus as measured by Enzyme-Linked Immunosorbent Assay (ELISA) between women vaccinated with BOOSTRIX or Td.
Time Frame: Pre-dose Day 1, One month after vaccination, at delivery, Day 180 (approximately 6 months after delivery)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 130 | 66
IU/mL
  Pre-vaccination | 1.3 [1.0 to 1.7] | 1.3 [0.9 to 1.9]
  One month after vaccination: number analyzed (Participants) | 129 | 66
  One month after vaccination | 6.6 [5.8 to 7.4] | 10.4 [8.8 to 12.2]
  Delivery: number analyzed (Participants) | 127 | 64
  Delivery | 3.3 [2.9 to 3.8] | 4.6 [3.9 to 5.5]
  6 months after delivery: number analyzed (Participants) | 65 | 35
  6 months after delivery | 2.9 [2.3 to 3.6] | 3.8 [3.1 to 4.5]
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for pre-vaccination time point; Test type: Superiority; p = 0.8370, t-test, 2 sided; Test compares difference in log values; Ratio = 1.0, 95% CI 2-sided [0.6 to 1.5] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for one month after vaccination time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 0.6, 95% CI 2-sided [0.5 to 0.8] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for delivery time point; Test type: Superiority; p = 0.0050, t-test, 2 sided; Test compares difference in log values; Ratio = 0.7, 95% CI 2-sided [0.6 to 0.9] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for 6 months after delivery time point; Test type: Superiority; p = 0.0689, t-test, 2 sided; Test compares difference in log values; Ratio = 0.8, 95% CI 2-sided [0.6 to 1.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

12. Secondary Outcome: GMC of Serum IgG Antibodies to Diphtheria in Pregnant Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to Diphtheria as measured by Enzyme-Linked Immunosorbent Assay (ELISA) between women vaccinated with BOOSTRIX or Td.
Time Frame: Pre-dose Day 1, One month after vaccination, at delivery, Day 180 (approximately 6 months after delivery)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Maternal | Td - Maternal
Number analyzed (Participants) | 130 | 66
IU/mL
  Pre-vaccination | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  One month after vaccination: number analyzed (Participants) | 129 | 66
  One month after vaccination | 1.3 [1.1 to 1.6] | 1.5 [1.1 to 2.0]
  Delivery: number analyzed (Participants) | 127 | 64
  Delivery | 0.8 [0.6 to 0.9] | 0.9 [0.6 to 1.2]
  6 months after delivery: number analyzed (Participants) | 65 | 33
  6 months after delivery | 0.6 [0.5 to 0.9] | 0.9 [0.6 to 1.4]
Statistical Analysis 1: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for pre-vaccination time point; Test type: Superiority; p = 0.8361, t-test, 2 sided; Test compares difference in log values; Ratio = 1.0, 95% CI 2-sided [0.7 to 1.6] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for one month after vaccination time point; Test type: Superiority; p = 0.5136, t-test, 2 sided; Test compares difference in log values; Ratio = 0.9, 95% CI 2-sided [0.6 to 1.3] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for delivery time point; Test type: Superiority; p = 0.4237, t-test, 2 sided; Test compares difference in log values; Ratio = 0.9, 95% CI 2-sided [0.6 to 1.2] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Maternal vs Td - Maternal; Statistical analysis for 6 months after delivery time point; Test type: Superiority; p = 0.1607, t-test, 2 sided; Test compares difference in log values; Ratio = 0.7, 95% CI 2-sided [0.4 to 1.2] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

13. Secondary Outcome: GMC of Serum IgG Antibodies to FHA in Infants Born to Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to FHA as measured by Enzyme-Linked Immunosorbent Assay (ELISA) at birth between infants born to women vaccinated with BOOSTRIX or Td.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 124 | 64
IU/mL
  At birth | 387.5 [327.9 to 457.9] | 28.4 [22.2 to 36.3]
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age): number analyzed (Participants) | 114 | 59
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age) | 143.5 [121.8 to 169.1] | 13.3 [10.1 to 17.6]
  One month after receipt of first dose of DTwP (approximately 10 weeks of age): number analyzed (Participants) | 58 | 32
  One month after receipt of first dose of DTwP (approximately 10 weeks of age) | 89.4 [70.7 to 113.2] | 8.7 [6.2 to 12.3]
  One month after receipt of last dose of DTwP (approximately 18 weeks of age): number analyzed (Participants) | 50 | 25
  One month after receipt of last dose of DTwP (approximately 18 weeks of age) | 46.2 [37.8 to 56.4] | 22.5 [15.9 to 31.7]
  6 months of age: number analyzed (Participants) | 63 | 32
  6 months of age | 23.9 [19.2 to 29.8] | 20.7 [14.2 to 30.2]
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for birth time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 13.7, 95% CI 2-sided [10.2 to 18.3] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for prior to receipt of first dose of DTwP (approximately 6 weeks of age); Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 10.8, 95% CI 2-sided [8.0 to 14.5] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of first dose of DTwP (approximately 10 weeks of age) time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 10.2, 95% CI 2-sided [6.9 to 15.2] — Difference in log values back transformed into ratio. Test compares difference in log values; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of last dose of DTwP (approximately 18 weeks of age) time point; Test type: Superiority; p = 0.0002, t-test, 2 sided; Test compares difference in log values; Ratio = 2.1, 95% CI 2-sided [1.4 to 3.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 5: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for 6 months of age time point; Test type: Superiority; p = 0.4828, t-test, 2 sided; Test compares difference in log values; Ratio = 1.2, 95% CI 2-sided [0.8 to 1.7] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

14. Secondary Outcome: GMC of Serum IgG Antibodies to PRN in Infants Born to Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to PRN as measured by Enzyme-Linked Immunosorbent Assay (ELISA) at birth between infants born to women vaccinated with BOOSTRIX or Td.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 124 | 64
IU/mL
  At birth | 184.5 [130.6 to 260.6] | 4.0 [2.7 to 5.9]
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age): number analyzed (Participants) | 114 | 59
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age) | 72.6 [51.7 to 101.9] | 1.8 [1.3 to 2.7]
  One month after receipt of first dose of DTwP (approximately 10 weeks of age): number analyzed (Participants) | 58 | 32
  One month after receipt of first dose of DTwP (approximately 10 weeks of age) | 47.1 [33.2 to 66.8] | 4.5 [3.1 to 6.6]
  One month after receipt of last dose of DTwP (approximately 18 weeks of age): number analyzed (Participants) | 50 | 25
  One month after receipt of last dose of DTwP (approximately 18 weeks of age) | 48.6 [34.9 to 67.8] | 80.2 [52.2 to 123.1]
  6 months of age: number analyzed (Participants) | 63 | 32
  6 months of age | 28.4 [21.6 to 37.3] | 39.1 [28.2 to 54.2]
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for birth time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 46.4, 95% CI 2-sided [26.6 to 81.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for prior to receipt of first dose of DTwP (approximately 6 weeks of age); Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 39.5, 95% CI 2-sided [24.0 to 65.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of first dose of DTwP (approximately 10 weeks of age) time point; Test type: Superiority; p < 0.0001, t-test, 2 sided; Test compares difference in log values; Ratio = 10.4, 95% CI 2-sided [6.1 to 17.9] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of last dose of DTwP (approximately 18 weeks of age) time point; Test type: Superiority; p = 0.0746, t-test, 2 sided; Test compares difference in log values; Ratio = 0.6, 95% CI 2-sided [0.3 to 1.1] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 5: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for 6 months of age time point; Test type: Superiority; p = 0.1532, t-test, 2 sided; Test compares difference in log values; Ratio = 0.7, 95% CI 2-sided [0.5 to 1.1] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

15. Secondary Outcome: GMC of Serum IgG Antibodies to Tetanus in Infants Born to Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to Tetanus as measured by Enzyme-Linked Immunosorbent Assay (ELISA) at birth between infants born to women vaccinated with BOOSTRIX or Td.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 124 | 64
IU/mL
  At birth | 4.1 [3.5 to 4.8] | 5.9 [5.0 to 7.0]
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age): number analyzed (Participants) | 114 | 59
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age) | 1.4 [1.2 to 1.6] | 2.0 [1.7 to 2.4]
  One month after receipt of first dose of DTwP (approximately 10 weeks of age): number analyzed (Participants) | 58 | 32
  One month after receipt of first dose of DTwP (approximately 10 weeks of age) | 0.8 [0.6 to 0.9] | 1.1 [0.9 to 1.3]
  One month after receipt of last dose of DTwP (approximately 18 weeks of age): number analyzed (Participants) | 50 | 25
  One month after receipt of last dose of DTwP (approximately 18 weeks of age) | 0.9 [0.6 to 1.2] | 1.5 [0.9 to 2.4]
  6 months of age: number analyzed (Participants) | 63 | 32
  6 months of age | 0.8 [0.6 to 1.1] | 1.0 [0.7 to 1.4]
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for birth time point; Test type: Superiority; p = 0.0022, t-test, 2 sided; Test compares difference in log values; Ratio = 0.7, 95% CI 2-sided [0.6 to 0.9] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for prior to receipt of first dose of DTwP (approximately 6 weeks of age); Test type: Superiority; p = 0.0008, t-test, 2 sided; Test compares difference in log values; Ratio = 0.7, 95% CI 2-sided [0.5 to 0.8] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of first dose of DTwP (approximately 10 weeks of age) time point; Test type: Superiority; p = 0.0261, t-test, 2 sided; Test compares difference in log values; Ratio = 0.7, 95% CI 2-sided [0.5 to 1.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of last dose of DTwP (approximately 18 weeks of age) time point; Test type: Superiority; p = 0.0532, t-test, 2 sided; Test compares difference in log values; Ratio = 0.6, 95% CI 2-sided [0.3 to 1.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 5: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for 6 months of age time point; Test type: Superiority; p = 0.5587, t-test, 2 sided; Test compares difference in log values; Ratio = 0.9, 95% CI 2-sided [0.5 to 1.4] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

16. Secondary Outcome: GMC of Serum IgG Antibodies to Diphtheria in Infants Born to Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to Diphtheria as measured by Enzyme-Linked Immunosorbent Assay (ELISA) at birth between infants born to women vaccinated with BOOSTRIX or Td.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 124 | 64
IU/mL
  At birth | 0.8 [0.7 to 1.0] | 0.9 [0.7 to 1.3]
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age): number analyzed (Participants) | 114 | 59
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age) | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4]
  One month after receipt of first dose of DTwP (approximately 10 weeks of age): number analyzed (Participants) | 58 | 32
  One month after receipt of first dose of DTwP (approximately 10 weeks of age) | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  One month after receipt of last dose of DTwP (approximately 18 weeks of age): number analyzed (Participants) | 50 | 25
  One month after receipt of last dose of DTwP (approximately 18 weeks of age) | 0.2 [0.2 to 0.3] | 0.4 [0.2 to 0.6]
  6 months of age: number analyzed (Participants) | 63 | 32
  6 months of age | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for birth time point; Test type: Superiority; p = 0.5056, t-test, 2 sided; Test compares difference in log values; Ratio = 0.9, 95% CI 2-sided [0.6 to 1.3] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for prior to receipt of first dose of DTwP (approximately 6 weeks of age); Test type: Superiority; p = 0.9466, t-test, 2 sided; Test compares difference in log values; Ratio = 1.0, 95% CI 2-sided [0.7 to 1.5] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of first dose of DTwP (approximately 10 weeks of age) time point; Test type: Superiority; p = 0.6911, t-test, 2 sided; Test compares difference in log values; Ratio = 1.1, 95% CI 2-sided [0.6 to 2.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of last dose of DTwP (approximately 18 weeks of age) time point; Test type: Superiority; p = 0.0952, t-test, 2 sided; Test compares difference in log values; Ratio = 0.6, 95% CI 2-sided [0.3 to 1.1] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 5: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for 6 months of age time point; Test type: Superiority; p = 0.4134, t-test, 2 sided; Test compares difference in log values; Ratio = 1.2, 95% CI 2-sided [0.8 to 2.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

17. Secondary Outcome: GMC of Serum IgG Antibodies to Fimbriae 2/3 (FIM 2/3) in Infants Born to Women Receiving BOOSTRIX or Td
Description: GMC of serum IgG antibodies to FIM 2/3 as measured by Enzyme-Linked Immunosorbent Assay (ELISA) at birth between infants born to women vaccinated with BOOSTRIX or Td.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 124 | 64
IU/mL
  At birth | 23.9 [17.8 to 32.0] | 15.2 [9.8 to 23.8]
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age): number analyzed (Participants) | 114 | 59
  Prior to receipt of first dose of DTwP (approximately 6 weeks of age) | 9.5 [7.1 to 12.7] | 6.9 [4.5 to 10.4]
  One month after receipt of first dose of DTwP (approximately 10 weeks of age): number analyzed (Participants) | 58 | 32
  One month after receipt of first dose of DTwP (approximately 10 weeks of age) | 10.9 [7.8 to 15.3] | 6.8 [4.8 to 9.7]
  One month after receipt of last dose of DTwP (approximately 18 weeks of age): number analyzed (Participants) | 50 | 25
  One month after receipt of last dose of DTwP (approximately 18 weeks of age) | 254.0 [153.3 to 420.6] | 517.6 [292.2 to 916.8]
  6 months of age: number analyzed (Participants) | 63 | 32
  6 months of age | 274.3 [191.7 to 392.6] | 465.6 [316.7 to 684.6]
Statistical Analysis 1: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for birth time point; Test type: Superiority; p = 0.0859, t-test, 2 sided; Test compares difference in log values; Ratio = 1.6, 95% CI 2-sided [0.9 to 2.6] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 2: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for prior to receipt of first dose of DTwP (approximately 6 weeks of age); Test type: Superiority; p = 0.2040, t-test, 2 sided; Test compares difference in log values; Ratio = 1.4, 95% CI 2-sided [0.8 to 2.3] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 3: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of first dose of DTwP (approximately 10 weeks of age) time point; Test type: Superiority; p = 0.0763, t-test, 2 sided; Test compares difference in log values; Ratio = 1.6, 95% CI 2-sided [1.0 to 2.7] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 4: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for one month after receipt of last dose of DTwP (approximately 18 weeks of age) time point; Test type: Superiority; p = 0.0836, t-test, 2 sided; Test compares difference in log values; Ratio = 0.5, 95% CI 2-sided [0.2 to 1.1] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group
Statistical Analysis 5: Comparison: BOOSTRIX - Infant vs Td - Infant; Statistical analysis for 6 months of age time point; Test type: Superiority; p = 0.0672, t-test, 2 sided; Test compares difference in log values; Ratio = 0.6, 95% CI 2-sided [0.3 to 1.0] — Difference in log values back transformed into ratio; The ratio is calculated as the GMC of the BOOSTRIX group divided by the GMC of the Td group

18. Secondary Outcome: Geometric Mean Ratio (GMR) of Maternal and Infant-specific Tdap-specific Antibodies
Description: GMR of maternal and infant-specific Tdap-specific antibodies (PT, FHA, PRN, tetanus, diphtheria) as measured by ELISA at delivery/birth after intrapartum receipt of BOOSTRIX versus Td. GMR represents the geometric mean ratio in infant antibody concentration at birth to maternal antibody concentration at delivery.
Time Frame: Time of delivery
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | BOOSTRIX - Infant | Td - Infant
Number analyzed (Participants) | 124 | 64
ratio
  Pertussis Toxin (PT) | 1.2 [1.1 to 1.2] | 0.8 [0.7 to 0.9]
  Filamentous Hemagluttin (FHA) | 1.2 [1.2 to 1.3] | 0.9 [0.8 to 1.0]
  Pertactin (PRN) | 1.1 [1.1 to 1.2] | 0.8 [0.7 to 0.9]
  Tetanus | 1.2 [1.2 to 1.3] | 1.3 [1.2 to 1.3]
  Diphtheria | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.1]

ADVERSE EVENTS:
Time Frame: Study vaccine-related Serious Adverse Events (SAE) occurring from the time of study vaccination through 6 months postpartum (180 days of life for the infant visit) for pregnant participants and infants were collected. Solicited Adverse Events (AEs) were collected from time of study vaccination through 7 days after study vaccination (Day 8). Unsolicited non-serious AEs were collected from time of study vaccination through approximately 30 days after study vaccination (Day 31).
Description: Total number of participants At Risk includes all maternal participants who received the study vaccine or infants born to mothers who received the study vaccine.
Arm/Group | BOOSTRIX - Maternal | Td - Maternal | BOOSTRIX - Infant | Td - Infant
All-Cause Mortality (participants affected / at risk) | 1/133 | 0/67 | 8/126 | 3/66
Serious Adverse Events (participants affected / at risk) | 20/133 | 10/67 | 13/126 | 6/66
Other Adverse Events (participants affected / at risk) | 35/133 | 24/67 | 0/126 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOOSTRIX - Maternal (N=133) | Td - Maternal (N=67) | BOOSTRIX - Infant (N=126) | Td - Infant (N=66)
Preterm Delivery (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Preterm Birth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 7 (7) | 4 (4)
Postpartum Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fetal Distress (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Imminent Uterine Rupture (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perinatal Anoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cleft Lip and Palate (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal Infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cephalopelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroplacental hematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prolong Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOOSTRIX - Maternal (N=133) | Td - Maternal (N=67) | BOOSTRIX - Infant (N=126) | Td - Infant (N=66)
Injection site pain (General disorders) | 9 (9) | 10 (10) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 20 (21) | 11 (12) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 7 (7) | 2 (3) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 10 (10) | 6 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03589768/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT03589768/SAP_002.pdf
  • Informed Consent Form (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03589768/ICF_000.pdf